CLINICAL TRIAL: NCT01506310
Title: Randomized Comparative Trial on the Efficacy of Behavioral Therapy, Exercise and Their Combination in Gestational Diabetes Mellitus (GDM).
Brief Title: Efficacy of Behavioral Therapy and Exercise in Gestational Diabetes Mellitus (GDM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, Principal Investigator, MD, Professor Assistant, Department of Internal Medicine, University of Turin, Italy
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: sbo2010
Record Dates: First submitted 2011-12-26; First posted 2012-01-10 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Birth-weight
Keywords: gestational diabetes mellitus; fasting glucose; insulin resistance; birth-weight; Glucose values; Insulin concentrations; Cesarean sections
MeSH Terms: conditions — Birth Weight; Diabetes, Gestational; Insulin Resistance | interventions — Behavior Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diet alone (No Intervention)
- Behavioral therapy (Experimental)
  Interventions: Behavioral: Behavioral therapy
- Exercise (Experimental)
  Interventions: Other: Exercise
- Behavioral therapy and exercise (Experimental)
  Interventions: Other: Behavioral therapy and exercise

INTERVENTIONS:
Behavioral: Behavioral therapy — General written dietary recommendations (about cooking, lowering sugar intake, reducing salt intake, reducing beverages and food with added sugars) and written options for dining out. A brief written guide on behavior change.
  Arms: Behavioral therapy
Other: Exercise — The exercise groups will be advised to walk at least 20-minute a day.
  Arms: Exercise
Other: Behavioral therapy and exercise — General written dietary recommendations (about cooking, lowering fat intake, reducing salt intake, reducing beverages and food with added sugars) and written options for dining out.
  Written recommendations for physical activity A brief written guide on behavior change
  Arms: Behavioral therapy and exercise

SUMMARY:
The purpose of the study is to test whether four lifestyle intervention programs (diet alone; diet and behavioral therapy, diet and exercise, diet and behavioral therapy and exercise), delivered to women with GDM during 24-26 weeks of gestational age will help women to improve their metabolic pattern, and decrease the incidence of adverse maternal and neonatal outcomes.

DETAILED DESCRIPTION:
Women with gestational diabetes (GDM) are at increased risk of adverse pregnancy and neonatal outcomes. It is estimated that most women diagnosed with GDM can achieve targeted glycemic goals with nutrition therapy alone. A moderate exercise is recommended to lower serum glucose and to improve insulin sensitivity. Despite this, few reports examine the effect of exercise on glucose intolerance during pregnancy. Furthermore, no trial on the efficacy of behavioral treatment in women with GDM is available.

The purpose of the study is to test whether four lifestyle intervention programs (diet alone; diet and behavioral therapy, diet and exercise, diet and behavioral therapy and exercise), delivered to women with GDM during 24-26 weeks of gestational age will help women to improve their metabolic pattern, and decrease the incidence of adverse maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 24 and 26 weeks
* Diagnosis of GDM at the 75g oral glucose tolerance test (OGTT)
* Singleton pregnancy

Exclusion Criteria:

* Body mass index > 40 or < 12kg/m2
* Any known diseases (pre-existing diabetes mellitus, cardiovascular diseases, liver/kidney diseases, cancers, arterial hypertension)
* Patients on any drugs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2009-07; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Serum fasting glucose values. | Fasting glucose will be measured at recruitment (24 weeks of gestation) and at the end of follow-up (38 weeks of gestation)
  To investigate changes from baseline in serum fasting glucose values in each arm with a 2x2 factorial design.

SECONDARY OUTCOMES:
Serum fasting insulin values | At recruitment (at 24 weeks of gestation) and at the end of follow-up (38 weeks of gestation)
  To investigate changes from baseline in serum fasting insulin values in each arm.
The need for insulin therapy | At recruitment and at the end of follow-up (38 weeks)
  The need for insulin therapy in each arm
The number of Cesarean sections | From recruitment until the date of delivery, either natural or by Caesarean section, assessed up to 42 weeks
  The number of Cesarean sections in each arm
The mean birth-weight of newborns | From recruitment until the date of delivery, assessed up to 42 weeks
  The mean birth-weight of newborns in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, Italy, Italy

REFERENCES:
- [Derived] Bo S, Gambino R, Menato G, Canil S, Ponzo V, Pinach S, Durazzo M, Ghigo E, Cassader M, Musso G. Isoleucine-to-methionine substitution at residue 148 variant of PNPLA3 gene and metabolic outcomes in gestational diabetes. Am J Clin Nutr. 2015 Feb;101(2):310-8. doi: 10.3945/ajcn.114.095125. Epub 2014 Dec 17. PMID 25646328
- See also: site for randomization — http://www.epiclin.it